CLINICAL TRIAL: NCT01789814
Title: The Effect of Prasugrel as Compared to Clopidogrel on Platelet Function Immediately Following the Termination of Intravenous Bivalirudin in Patients Undergoing Percutaneous Coronary and Structural Cardiac Intervention
Brief Title: Effect of Prasugrel Versus Clopidogrel on Platelet Function After Bivalirudin Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PraCloBiv2013CK; TMCcardintervCK2013 (Other: Tufts Medical Center)
Record Dates: First submitted 2013-02-04; First posted 2013-02-12 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous Coronary Intervention; Platelet Aggregation Inhibitors; bivalirudin
MeSH Terms: conditions — Coronary Artery Disease | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Active Comparator): Prasugrel oral loading dose of 60 mg administered preceding cardiac intervention
  Interventions: Drug: Prasugrel
- Clopidogrel (Active Comparator): Clopidogrel oral loading dose of 600 mg administered preceding cardiac intervention
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Prasugrel — Patients will be randomized to prasugrel or clopidogrel to assess the effect of these drugs on inhibition of platelet aggregation following the cessation of bivalirudin therapy.
  Other Names: Effient
  Arms: Prasugrel
Drug: Clopidogrel — Clopidogrel 600 mg as a loading dose immediately prior to the start of procedure and 75 mg daily thereafter
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
Early stent thrombosis has been noted with increased frequency in acute coronary syndrome (ACS) patients undergoing percutaneous coronary intervention (PCI) who are treated with bivalirudin and clopidogrel. The brief half life of bivalirudin acting in concert with the delayed action of clopidogrel likely exposes patients to thrombosis during a vulnerable period of reduced antiplatelet effect in the immediate post stenting period. Combination therapy with bivalirudin and prasugrel is conceptually attractive as the more rapid onset of action of prasugrel could potentially significantly diminish the vulnerable period, likely reducing the potential for acute stent thrombosis. The trials which have documented the efficacy of prasugrel as compared to clopidogrel have, in general, not reported on patients in whom bivalirudin was utilized. Currently, in the United States, bivalirudin is the most commonly used adjunctive agent used during PCI. Using light transmission aggregometry, this study will examine the inhibition of platelet aggregation in patients randomized to treatment with clopidogrel vs prasugrel during the vulnerable period following the discontinuation of bivalirudin therapy. The investigators anticipate that this study will document significant enhancement of inhibition of platelet aggregation in patients randomized to prasugrel treatment.

DETAILED DESCRIPTION:
Percutaneous coronary intervention (PCI) targeting coronary lesions in patients with coronary syndromes leads to iatrogenic endothelial disruption and heightened platelet activation and aggregation. Blocking platelet aggregation with glycoprotein (GP) IIb/IIIa inhibitors has been demonstrated to be of unequivocal benefit when combined with heparin in patients undergoing PCI. Heparin-mediated thrombin inhibition is an established therapy for safely performing PCI, however, there are several well known limitations of heparin including its variable anticoagulant effect due to nonlinear pharmacokinetics and inconsistent binding to blood proteins. In addition, heparin does not effectively block clot-bound thrombin and may cause thrombocytopenia.

The direct thrombin inhibitor (DTI), bivalirudin, which binds with high affinity to exosite I of thrombin, may be a safer alternative to other commonly used pharmacologic PCI adjuncts with an expert consensus document defining it as "reasonable to use as an alternative to unfractionated heparin and GP IIb/IIIa antagonists in low-risk patients undergoing elective PCI". The ACUITY trial has supported the use of bivalirudin in patients with unstable coronary syndromes. This study showed similar rates of ischemic events and less bleeding when compared with patients treated with heparin and GP IIb/IIIa inhibitors. Similar results were reported in the REPLACE-2 randomized trial, which studied a patient population with a lower prevalence of acute coronary syndromes. Recent results from our laboratory suggest that at least a part of the salutary effects of DTIs are due to a reduction of thrombin and to a lesser extent, collagen-mediated platelet activation.

Inhibition of the platelet P2Y12 Adenosine Diphosphate (ADP) receptor is standard of care when added to aspirin in patients undergoing coronary stenting. A 600 mg loading dose of clopidogrel led to enhanced inhibition of platelet aggregation and a reduction in adverse clinical outcomes in Non-ST-Segment Elevation Myocardial Infarction (NSTEMI) patients undergoing coronary stenting when compared to 300 mg. Other studies have documented that when compared with both 300 and 600 mg loading doses of clopidogrel, a 60 mg loading dose of prasugrel has been documented to eventuate in faster onset, greater magnitude and more consistent levels of platelet inhibition as measured by light transmission aggregometry. Several studies have documented significantly greater platelet inhibition with prasugrel treatment when compared to high-dose clopidogrel therapy. The more potent P2Y12 ADP receptor antagonist prasugrel significantly reduced the composite endpoint of cardiovascular death, nonfatal MI, and nonfatal stroke in higher-risk ACS patients referred for PCI. The salutary effects referable to prasugrel treatment in this study were mostly due to a reduction in the incidence of myocardial infarction.

In the HORIZONS AMI trial patients with ST-segment elevation myocardial infarction who underwent primary PCI, anticoagulation with bivalirudin alone, as compared with heparin plus GP IIb/IIIa inhibitors, resulted in significantly reduced 30-day rates of major bleeding and net adverse clinical events. Despite these results and those from our laboratory documenting a profound bivalirudin-mediated effect on platelet aggregation, closer analysis of the HORIZONS AMI trial has documented a higher acute stent thrombosis rate in bivalirudin as opposed to GP IIb/IIIa inhibitor treated patients. The investigators have recently documented that the half life of bivalirudin, at the currently utilized dose during cardiac interventions is 29.3 minutes. The relatively short half life of this DTI in concert with the relatively long time period required to activate clopidogrel from a prodrug to its active metabolite, likely exposes patients to a vulnerable period when there is suboptimal platelet inhibition. It is plausible that this vulnerable period when platelet activity is not inhibited was the proximate cause of early stent thrombosis in the HORIZONS trial. Consequently, earlier acting, more potent thienopyridine therapy, i.e. prasugrel, when combined with bivalirudin treatment has the potential to reduce bleeding (compared with GP IIb/IIIa inhibitors) while preventing peri-procedural MI as well as providing protection from platelet-mediated stent thrombosis (compared with clopidogrel) during the vulnerable period following PCI.

The overwhelming majority of published data examining clinical outcomes or in-vivo pharmacodynamic and pharmacokinetic differences between clopidogrel and prasugrel have done so in PCI patients in whom bivalirudin was either not used or used very infrequently, i.e. in less than 10% of studied patients. However, at the present time in the United States, bivalirudin is the preeminent antithrombotic adjunctive therapy used during PCI. Consequently, comparative data regarding the effect of prasugrel and clopidogrel on platelet function in bivalirudin-treated patients is of significant clinical importance.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent before initiation of any study related procedures
2. Male or non-pregnant female aged 18 to ≤ 75 years
3. Referred for PCI or structural cardiac intervention and planned to receive bivalirudin treatment
4. Only subjects in whom the treating physician feels that clopidogrel and prasugrel are equivalent on the basis of available clinical literature will be included.

Exclusion Criteria:

1. Currently receiving glycoprotein IIb/IIIa inhibitors.
2. Have received prasugrel or clopidogrel within 2 weeks
3. Serum creatinine level >2.0
4. Hypersensitivity to bivalirudin, prasugrel, clopidogrel or aspirin
5. Currently on heparin administration or administered ≤ 4.5 h prior to intervention
6. Thrombocytopenia (<50,000/µL)
7. Severe systemic hypertension defined as systolic blood pressure >180 mm Hg and/or diastolic blood pressure >110 mm Hg
8. Body weight < 60 kg
9. Cardiogenic shock
10. Acute pericarditis
11. Active internal bleeding
12. History of bleeding diathesis within previous thirty days
13. Any history of intracranial hemorrhage, Transient ischemic attack (TIA ) or stroke
14. Arteriovenous malformations or aneurysms
15. Major surgical procedures or severe physical trauma within last thirty days.
16. Symptoms or findings suggestive of aortic dissection
17. Pregnancy
18. Participation in other clinical research studies involving the evaluation of investigational drugs or devices within 30 days of enrollment
19. Incompetent subjects or subjects otherwise unable to provide informed consent
20. Subjects in whom the treating physician believes that one agent (prasugrel or clopidogrel) is preferable over the other will be excluded from study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carey Kimmelstiel, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 24 subjects were enrolled to complete this study. The enrollment process took place in the adult cardiac catheterization laboratory at this hosptial. The inform consent process took place at the subject arrival time for the date procedure.
Pre-assignment Details: The randomized arm assignment was done by numbered envelopes. Once it was confirmed the subject was going to have a coronary intervention, the correspondent envelope was opened to assign the study arm drug.
Period: Overall Study
Arm/Group | Prasugrel | Clopidogrel
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Clopidogrel | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.41 (9.80) | 62.5 (80.5) | 61.99 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 11 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 11 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in ADP-mediated Platelet Aggregation, APP, SFFLRN, AYPGKF.
Description: To document the extent of inhibition of ADP mediated platelet aggregation following the discontinuation of bivalirudin therapy in patients treated with prasugrel as compared to patients treated with clopidogrel.
  The percent inhibition of platelet aggregation was measured by light transmission aggregometry of platelet-rich plasma in response to P2Y12 and PAR1 and PAR4 thrombin receptor agonists at baseline and at 1, 2, 4 and 16 h following the cessation of bivalirudin infusion. Platelet response to agonists: 20 mM ADP(P2Y12), 5 mM SFLLRN (PAR1), and 160 mM AYPGKF (PAR4) was performed. The magnitude of inhibition of platelet aggregation for each agonist was calculated as the mean final change from baseline in light transmission aggregometry at each time point.
Time Frame: Baseline, 60, 120, 240, 960 mins following termination of bivalirudin infusion
Population: 24 patients referred for intervention with planned bivalirudin therapy, not previously treated with a P2Y12 inhibitor and not receiving heparins or GP IIb/IIIa inhibitors were randomized to treatment with either clopidogrel (600 mg) or prasugrel (60 mg).
Measure: Number; unit: % inhibitn of platelet aggregation
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 12 | 12
% inhibitn of platelet aggregation
  ADP 20 uM-1 hour % | 84 | 38
  ADP 20 uM-2 hour % | 94 | 53
  ADP 20 uM-4 hour % | 98 | 85
  ADP 20 uM-16 hour % | 98 | 85
  SFFLRN 5 uM-1 hour | 62 | 2
  SFFLRN 5 uM-2 hour | 64 | 9
  SFFLRN 5 uM-4 hour | 75 | 17
  SFFLRN 5 uM-16 hour | 58 | 15
  AYP 160 uM-1 hour | 39 | 7
  AYP 160 uM-2 hour | 44 | 9
  AYP 160 uM-4 hour | 53 | 13
  AYP 160 uM-16 hour | 41 | 11
Statistical Analysis 1: Comparison: Prasugrel vs Clopidogrel; Each patient will have paired samples representing their baseline as well as an on-drug sample. The magnitude of platelet inhibition for each studied agonist will be performed utilizing mean maximal change from baseline in light transmission aggregometry. The paired samples will be analyzed using a two-tailed student's t-test. Statistical significance will be assumed to occur when p<0.05; Test type: Superiority or Other; p = 0.001, t-test, 2 sided — Prasugrel treatment when compared to Clopidogrel was associated with significant reduction in platelets aggregation for all plateles agonist (ADD, SFFFLRN, AYPGKF) at all measured time points

ADVERSE EVENTS:
Time Frame: Periprocedural period up to 24 hours
Arm/Group | Prasugrel | Clopidogrel
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No